CLINICAL TRIAL: NCT05808907
Title: Assessing Discrepancies in Patient/Physician Evaluation of Transcatheter Aortic Valve Implantation and Developing a Patients Reported Outcomes Based Model to Predict Procedure Benefits Using a Novel Patient-oriented Questionnaire
Brief Title: Patient Reported Outcomes (PROMs) in Transcatheter Aortic Valve Implantation (TAVI) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 453-18-RMC
Record Dates: First submitted 2018-07-08; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: PROM; Patient Reported Outcomes; Transcatheter Aortic Valve Implantation
Keywords: PROM; Patient reported outcomes; Transcatheter Aortic Valve Implantation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A novel TAVI PROMs questionnaire will be created by us and used for this study.

SUMMARY:
The transcatheter Aortic Valve Implantation (TAVI) population with severe aortic stenosis (AS) is characterized by advanced age (most patients are octogenarians) and multiple comorbidities. For elderly patients, improvements in heart failure symptoms, functional status, and quality of life (QOL) maybe as important as longevity or even more. Over the last decade, we observe a change in trend, estimating medical interventions by clinical parameters along with other non-clinical parameters indicating a day-to-day improvement in factors which are more valuable to the patient and their families. This change is based on the understanding that treating a patient's physical symptoms successfully does not necessarily mean improving their QOL. The patient reported outcome measures (PROMs) initiative is focused upon what matters to patients during and following medical interventions. Data on PROMs in TAVI patients is increasing over the years but is still lacking, despite its potential to improve patient's care. In this study, we intend to create a novel self-developed patient-oriented PROM questionnaire specifically for TAVI patients and use it to assess the differences between physician's and patient's perception of a successful TAVI procedure. These discrepancies will form the basis for building a forecast model for a successful TAVI from the patient's perspective.

DETAILED DESCRIPTION:
The transcatheter Aortic Valve Implantation (TAVI) population with severe aortic stenosis (AS) is characterized by advanced age (most patients are octogenarians) and multiple comorbidities. For elderly patients, improvements in heart failure symptoms, functional status, and quality of life (QOL) maybe as important as longevity or even more. Over the last decade, we observe a change in trend, estimating medical interventions by clinical parameters along with other non-clinical parameters indicating a day-to-day improvement in factors which are more valuable to the patient and their families. This change is based on the understanding that treating a patient's physical symptoms successfully does not necessarily mean improving their QOL. The patient reported outcome measures (PROMs) initiative is focused upon what matters to patients during and following medical interventions. A Patient Reported Outcome (PRO) is "any report of the status of a patient's health condition that comes directly from the patient, without interpretation of the patient response by a clinician or anyone else". Data on PROMs in TAVI patients is increasing over the years but is still lacking, despite its potential to improve patient's care. Until recently, studies have used pre-validated questionnaires (such as KCCQ, ED-5D, PROMIS-10 or SF-36) for other patient's populations and validated them for the TAVI patient's population. Recently, the MacNew questionnaire was validated for TAVI patients. However, as far as we know, no questionnaire has been developed in collaboration with TAVI patients. As we believe that patient's involvement in a PROM's development is essential to truly capture patient's perspective, we decided to develop a new questionnaire collaborating with TAVI patients instead of using a pre-validated questionnaire.

In this research proposal our main objective is to define what is a successful TAVI in the patient's perspective. To do so, we wish to create and validate a new TAVI PROM questionnaire RT-20 (Rabin TAVI 20 questions questionnaire) and use it to assess the differences between physician's and patient's perception of a successful TAVI procedure. In the first phase, to form the questionnaire, 30 patients up to 6 months after TAVI procedure, will be recruited to choose the questions from a questions' repository. To validate the questionnaire, 30 physicians (cardiology consultants, internal medicine, and geriatrics consultants) will be recruited to assure content validity and 30 new patients after TAVI will be recruited to examine the face validity of the questionnaire. In the second phase, after obtaining the validated RT-20 questionnaire, 150 new patients will be recruited for the two discrepancies assessments: the first, between patient's perception and his/her physician's perception and the second, between physician himself before and after exposure to the RT-20 validated questionnaire regarding the successfulness of the TAVI procedure. All patients and physicians will be recruited from Rabin Medical Center - Beilinson campus.

These discrepancies will form the basis for building a forecast model for a successful TAVI from the patient's perspective. We will look for independent predictors of disagreement between patients and physicians as to the success of the procedure; as well as predictors of the physician's assessment before and after seeing the PROM questionnaire RT-20. These possible determinants such as living alone, need for assistance in activities of daily living and multiple comorbidities will be entered into a logistic regression model. We will also build a model to predict the patient satisfaction with the procedure. This model will help to aid in the triage of patients suffering from severe AS in an attempt to avoid futile procedures and thus optimize procedural success and/or resources utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (men and women) who underwent a successful TAVI procedure (defined according to VARC 2) REF
2. Patients who agreed to participate in the study and gave their written inform consent.
3. Patients who are capable to fulfill the PROMs questionnaires.

Exclusion Criteria:

1. Patients that are not able to give their consent.
2. Patients that from any reason are not able to fulfill the PROM's questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Transcatheter Aortic Valve Implantation (TAVI) Patients before and after the procedure
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-09-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Dependent variable (model) - Successful TAVI from the patient perspective. | Before the TAVI procedure until 3 months after it.
  In this research our main objective is to define what is a successful TAVI in the patient's perspective. To do so, we will create and validate a new TAVI PROM questionnaire RT-20 (Rabin TAVI 20 questions questionnaire) and use it to assess the differences between physician's and patient's perception of a successful TAVI procedure. These differences will be used to build a model to predict the patient satisfaction with the TAVI procedure. This model will help to aid in the triage of patients suffering from severe AS in an attempt to avoid futile procedures and thus optimize procedural success and/or resources utilization.
The disagreement between the patient and his/her doctor's perception | Before the TAVI procedure until 3 months after it.
  For the discrepancy assessment part, the following outcomes will be measured: Primary - The disagreement between the patient and his/her doctor's perception of the patient's health, measured at 3 months FU visit by the Likert scale.
correlation assessment between patient's survival and patient's RT-20 score | Before the TAVI procedure until 12months after it.
  For the correlation assessment between patient's survival and patient's RT-20 score part: Primary outcome - Correlation extent between patient's survival 12 months post TAVI and patient's RT-20 score.

SECONDARY OUTCOMES:
The disagreement between the doctor's perception before and after observing the RT-20 questionnaire. | Before the TAVI procedure until 3 months after it.
  For the discrepancy assessment part, the following outcomes will be measured: Secondary outcome - The disagreement between the doctor's perception (regarding the successfulness of the TAVI) before and after the exposure to the RT-20 questionnaire (representing the patient's perception of his health status and the successfulness of the TAVI procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Ran Kornowski, MD FESC FACC, Study Chair — Chairmain of Cardiology devision
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel